CLINICAL TRIAL: NCT04639570
Title: KneuroKnits: Evaluating Social Participation and Anxiety Response Associated With Participation in a Knitting Group for People With Neurological Conditions (Pilot Study)
Brief Title: KneuroKnits: Participation and Anxiety in People With Neurological Conditions Participating in a Knitting Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-717
Record Dates: First submitted 2020-11-02; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders; Acquired Brain Injury; Physical Disability
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KneuroKnits group (Experimental): Participants in the KneuroKnits group
  Interventions: Other: KneuroKnits

INTERVENTIONS:
Other: KneuroKnits — The KneuroKnits program will be based upon current knitting education practices and leading practices in facilitation of social participation for individuals with neurodevelopmental disorders, physical disabilities, and acquired brain injuries. The program will consist of 4 weekly sessions in which participants will learn knitting fundamentals and have opportunities to socialize over a shared occupation. The 4 weekly sessions of the KneuroKnits curriculum will include related knitting and social skills themes of the week. Each session will begin with a structured lesson on the knitting topic of the day, and will then continue into knitting practice and social interaction. Participants will be encouraged to practice their new skills (knitting and social) between sessions, and will be allowed to keep all materials that they use or create.

SUMMARY:
The reported social benefits of knitting combined with the urgent need for social and activity-based programs in the disability community suggest that a knitting intervention may fill a substantial gap in available programs. Knitting may also be well suited to autistic strengths, combining sensory aspects (colourful sights, soft touch, rhythmic sounds), visual patterning, and repetitive actions. Surprisingly, no knitting programs for ASD or other conditions are reported in the literature. It is proposed that a knitting group can provide social and skill-building opportunities, improving real-world social outcomes for youth with ASD, and resulting in KneuroKnits, a program designed specifically to serve this need. The program will be designed and run by a collaborative team of clinicians, researchers, knitting experts, and a self-advocate with ASD. This program will enhance evidence supporting programs providing contexts for the dual goals of meaningful social interaction for young people with neurodevelopmental disorders, physical disabilities, and acquired brain injuries and building a real world creative skill that can facilitate social interaction within and beyond the program. This study will evaluate participants' experiences of the program as well as their levels of anxiety at various points during the program.

DETAILED DESCRIPTION:
This study has two sets of aims. The first are related to social and environmental experiences, and the second are related to anxiety experiences.

Aim 1: Social and environmental experiences

1. To qualitatively observe and understand the social and skill-building experiences of a knitting group for people with neurodevelopmental disorders, physical disabilities, and acquired brain injuries from the perspectives of participants, their parents, and program facilitators;
2. To explore whether a professionally facilitated knitting group is perceived to be a beneficial and/or enjoyable environment for people with neurodevelopmental disorders, physical disabilities, and acquired brain injuries to socialize with peers;
3. To explore whether a professionally facilitated knitting group is perceived as an appropriate and/or desired learning or skill building environment for people with neurodevelopmental disorders, physical disabilities, and acquired brain injuries; and
4. To collect data that will drive the creation of a manualized KneuroKnits program and funding for future quantitative outcome measurements of program success.

Aim 2: Anxiety

a. To evaluate the impact of a knitting instructional program on self report of anxiety in individuals with neurodevelopmental disorders, physical disabilities, and/or acquired brain injuries.

Program design:

The KneuroKnits program will be based upon current knitting education practices and leading practices in facilitation of social participation for youth with neurodevelopmental disorders, physical disabilities, and acquired brain injuries. The program will consist of 4 weekly sessions in which participants will learn knitting fundamentals and have opportunities to socialize over a shared occupation. The 4 weekly sessions of the KneuroKnits curriculum will include related knitting and social skills themes of the week. Each session will begin with a structured lesson on the knitting topic of the day, and will then continue into knitting practice and social interaction. Participants will be encouraged to practice their new skills (knitting and social) between sessions, and will be allowed to keep all materials that they use or create. The project involves two pilot runs of the program in a pre-post study design.

Research Design:

The research includes both qualitative and quantitative components, all of which align with the structure of the KneuroKnits program described above. The project has two complementary foci that will be evaluated separately: (1) social and skill based experiences of program participation, and (2) the impact of program participation on anxiety related responses.

1. Social and skill based experiences of program participation:

   Primarily using qualitative design driven by an interpretive phenomenological methodology, this study will explore program experiences using observation and interviews with participants and stakeholders. The research team will also evaluate the program environment (activity setting) using a validated measure (SEAS).
2. The impact of program participation on anxiety related responses:

This study will employ a pre-post design. Anxiety will be measured at 2 time points for all participants (baseline, week 4) using self report (the anxiety subscale of the Symptom Checklist 90 [SCL-90] and the State-Trait Anxiety Inventory [STAI] will be collected when the participant attends the relevant KneuroKnits session. If the participant misses that particular session, they will be asked to come in to Holland Bloorview at their earliest convenient time to complete the measures.

The program will be administered at two different sites to increase access to a broad population. In October-November 2018, the 4-week program will be conducted at the Ontario Science Centre site, and in November-December 2018, the program will be conducted at the Holland Bloorview site.

ELIGIBILITY:
Inclusion Criteria:

1. a confirmed diagnosis of a neurodevelopmental disorder, physical disability, and/or acquired brain injury;
2. no diagnosis of intellectual disability (IQ>=70);
3. aged 15-24;
4. can understand and follow single- or multi-step instructions with or without assistance (determined by personal or parental report); and
5. can manipulate knitting materials (yarn, needles) as they are or with modifications and/or assistance. Indicators of ability will include tasks such as ability to tie a shoe or button shirt buttons.

Exclusion Criteria:

1) has engaged in self-harm or physical aggression in the past 6 months, due to safety risks with knitting needles

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2018-11-03 (Actual); Primary Completion 2019-02-09 (Actual); Study Completion 2019-02-09 (Actual)

PRIMARY OUTCOMES:
Self-reported Experience of Activity Settings (SEAS) | End of first session (week 1)
  The SEAS is a validated measure of participants' self-reports of their experiences of activity settings.
Self-reported Experience of Activity Settings (SEAS) | End of last session (week 4)
  The SEAS is a validated measure of participants' self-reports of their experiences of activity settings.
Symptom Checklist-90 (SCL-90; anxiety subscale; change during program participation) | Week 1
  The SCL-90 has been used to evaluate anxiety in adults with ASD and is a broadly used measure in adults.
Symptom Checklist-90 (SCL-90; anxiety subscale; change during program participation) | Week 4
  The SCL-90 has been used to evaluate anxiety in adults with ASD and is a broadly used measure in adults.
State-Trait Anxiety Inventory (STAI; change between beginning and end of sessions; change between weeks 1 and 4) | Beginning of Session 1 (week 1)
  Measure of current symptoms of anxiety.
State-Trait Anxiety Inventory (STAI; change between beginning and end of sessions; change between weeks 1 and 4) | End of Session 1 (week 1)
  Measure of current symptoms of anxiety.
State-Trait Anxiety Inventory (STAI; change between beginning and end of sessions; change between weeks 1 and 4) | Beginning of Session 4 (week 4)
  Measure of current symptoms of anxiety.
State-Trait Anxiety Inventory (STAI; change between beginning and end of sessions; change between weeks 1 and 4) | End of Session 4 (week 4)
  Measure of current symptoms of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Penner, MD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data may be shared upon reasonable request.